CLINICAL TRIAL: NCT03184922
Title: A Prospective, Randomised Study Investigating the Use of a Fixed Loop Versus an Adjustable Suspensory Loop in Anterior Cruciate Ligament Reconstruction - a Comparison of Clinical and Functional Outcome
Brief Title: Fixed Versus Adjustable Loop in ACL Reconstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1711539
Record Dates: First submitted 2017-05-24; First posted 2017-06-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: femoral suspensory loops

STUDY DESIGN:
Intervention Model Description: This is a blinded randomised controlled trial with 1 arm of the study having femoral side cortical fixation using a fixed length suspensory loop and the other an adjustable loop
Who Masked: Participant, Outcomes Assessor
Masking Description: 1. The patients will be informed they will not be told which arm of the study they are allocated to.
  2. The outcomes assessor for the KT1000 will be a physiotherapist not a surgeon and will not be told which type of surgery the patient has undergone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed suspensory loop (Active Comparator): Non-adjustable femoral cortical fixation device to be used
  Interventions: Procedure: Adjustable versus fixed suspensory loop femoral side graft fixation
- Adjustable suspensory loop (Experimental): Adjustable femoral cortical fixation device to be used
  Interventions: Procedure: Adjustable versus fixed suspensory loop femoral side graft fixation

INTERVENTIONS:
Procedure: Adjustable versus fixed suspensory loop femoral side graft fixation — A comparison of 2 different types of surgical technique for attaching the femoral side graft in ACL reconstruction: with a fixed suspensory loop or an adjustable one

SUMMARY:
Study Aims and Objectives:

To investigate the following null hypothesis: that there is no difference in clinical and functional outcome when comparing outcomes of Anterior Cruciate Ligament (ACL) reconstruction when comparing femoral side graft fixation with either a fixed versus an adjustable suspensory loop system.

The research team will achieve this aim by:

* Enrolling 150 patients into this study over a period of 2 years and 8 months
* Carrying out a prospective randomised study looking at the subject matter over a period of 5 years and 8 months
* Analysing patients functional status pre and post-surgery using patient generated questionnaires
* Quantitatively measuring knee joint laxity using the KT1000 testing device at the 3, 6 and 12 month post-surgery time frames
* Collating the data received into a spread sheet for analysis by a professional statistician.

It is not uncommon to tear the anterior cruciate ligament (ACL) particularly during sporting activities. Younger and sportier patients will often have this ligament reconstructed so as to allow them to return to sport with a stable knee joint that they feel they can trust.

Various surgical techniques exist to perform ACL reconstruction. In Exeter, the favoured technique is to reconstruct the ligament by taking two of the hamstring tendons from the back of the knee and creating a graft with these, passing them through a bony tunnel to replace the torn ACL. On the shin bone side of the knee the graft is fixed in place using a screw. On the thigh bone side, the graft is attached to a device known as a suspensory loop.

The length of the graft and the length of the tunnel in the thigh bone vary from patient to patient. It is important to get a good length of the graft material in both the shin and thigh bones so as to give the best chance of the graft attaching to the surrounding bone. With the fixed loop system, once the metal button attached to the outer thigh bone is in place, the length of the loop cannot be adjusted. Thus the amount of hamstring graft in either end of the bony tunnel cannot be changed. One potential advantage of an adjustable loop system is that the amount of graft in either end of the bone tunnel can be altered to ensure sufficient graft is accurately placed.

The research team are planning to run this study to identify which type of loop system gives the best outcome for patients, examining the results in different ways including questionnaires to measure how well the patients feel their knee is performing, and specific tests to measure knee function.

If patients consent to be in the study, they will be randomly allocated to receive one of the 2 ACL reconstruction options above and their progress monitored for 2 years after the operation. All aspects of surgical care will be as routine practice apart from the decision to fix the graft to the thigh bone with an adjustable or fixed suspensory loop.

DETAILED DESCRIPTION:
Research Question:

In the treatment of patients requiring anterior cruciate ligament (ACL) reconstruction, is there any difference in clinical and functional outcomes for patients when comparing femoral side graft fixation using a fixed loop versus an adjustable suspensory loop system?

Study Aims and Objectives:

1. To investigate the following null hypothesis: that there is no difference in clinical and functional outcome when comparing outcomes of ACL reconstruction when comparing the use of a fixed versus an adjustable suspensory loop system.
2. To identify the optimal surgical technique for patients requiring ACL reconstruction surgery.

The research team will achieve these aims by:

* Enrolling 150 patients into this study over a period of 2 years and 8 months
* Carrying out a prospective randomised study looking at the subject matter over a period of 5 years and 8 months
* Analysing patients functional status pre and post-surgery using patient generated questionnaires
* Quantitatively measuring knee joint laxity using the KT1000 testing device at the 3, 6 and 12 month post-surgery time frames
* Collating the data received into a spread sheet for analysis by a professional statistician

Background:

ACL rupture is a common injury. The National Ligament Registry (NLR) report (2016) details that 2585 patients with this injury were added to the Registry between 31/01/15 and 31/01/16. Of these, 1851 (71.6%) underwent reconstruction surgery and 734 patients (28.4%) were treated non-operatively. There is no clear consensus as to the best surgical technique for this procedure. However, one of the commonest techniques used is that involving the use of hamstring autograft- 95% of ACL reconstructions in Sweden in 2012 were performed using this method and 88% in the UK in 2015. A tunnel is drilled through the distal femur and proximal tibia, and the ACL graft passed through the tunnel. With this hamstring autograft method, various methods exist for fixing the graft on the femoral side- interference screws, transfemoral suspensory devices and femoral suspensory devices. There is no consensus as to which is best.

Rehabilitation after this type of surgery has become more aggressive over the years with early full weight-bearing, range of motion and strengthening exercises beginning soon after surgery. It is essential to preserve the initial stability of the graft whilst healing of the graft to the surrounding bony tunnel occurs so as to provide maximal benefit from the surgery for the patients. This healing process can take up to 12 weeks.

Failure of an ACL reconstruction can take different forms with graft stretching, graft failing to incorporate, traumatic re-rupture and infection being the most frequent causes. The assessment of ACL reconstruction failure can be performed in different ways. Samitier et al report the knee may demonstrate objective laxity (as tested by clinical tests such as Lachman and Pivot Shift or mechanical tests such as the KT1000). There may be a patient perception of instability even though objective tests are satisfactory). Using the KT1000 arthrometer, Alford and Bach report the rationale for a maximum manual side-to-side difference of 3 mm when assessing anterior tibial translation or an absolute laxity of 10 mm in the injured knee as the diagnostic criteria for ACL deficiency. Patient recorded outcome measures such as the Knee Osteo-arthritis Outcome Score (KOOS), Tegner activity scale and the International Knee Documentation Committee (IKDC) subjective questionnaire are all validated and can be used to assess satisfaction with surgical outcome and functional ability.

Suspensory fixation devices are used to draw the graft in to the femoral tunnel. Tunnel lengths differ between patients as do graft lengths. With a fixed length suspensory loop, once the metal device to fix the graft in the femoral tunnel has been deployed, it cannot be adjusted. In theory, fixed length suspensory loops may result in insufficient graft in the femoral tunnel. Whilst fixed suspensory loops are available in a multitude of sizes to overcome this problem, this will necessitate keeping a large stock of differing size products available in the operating theatre which will incur cost repercussions. With an adjustable suspensory loop, the graft can continue to be pulled up into the femoral tunnel even after the fixation button is attached to the outer femoral cortex giving the operating surgeon greater intra-operative flexibility. This will allow a greater amount of graft to be drawn within the femur. If one can have a short length of suspensory loop and a greater amount of graft in the tunnel, there will be less motion of the graft in the tunnel and a greater ability of the graft to unite to the surrounding bone.

If the harvested graft is unexpectedly found to be short, the adjustable loop may offer a further advantage to the surgeon over the fixed loop. In this situation, if the fixed loop is deployed, there may be a sub-optimal amount of graft in the tibial tunnel. Thus, there is less graft for the interference screw to engage against for fixation on the tibial side. In these circumstances, the ability for the surgeon to lengthen the loop, and pull some extra graft into the tibia will allow for better fixation of the graft on the tibial side.

Presently, the fixed loop devices are available in varying sizes. Keeping a range of different sized products in stock to cover graft length issues, will incur extra costs. A benefit of an adjustable loop system may be therefore, that it will only require the single size product to be kept on the shelf, with an implication for cost savings in terms of amount of stock that needs to be on hand.

There have been several biomechanical studies comparing the strength and lengthening of fixed versus suspensory loop devices in a laboratory environment. In particular, assessment is made of the lengthening of the suspensory loop when subject to repetitive cyclic loading and also of ultimate failure when subject to load to failure testing. Varying results have been reported. Petre et al showed 4 suspensory loops had ultimate failure tolerances that would exceed the forces that an ACL graft would be subjected to. However, on repetitive cyclic testing one of the adjustable length suspensory loops stretched in excess of 3mm which was beyond the threshold which would be considered a clinical failure.

Eguchi et al reported a fixed loop suspensory device as having greater statistically significant strength and lower total displacement/ stretching values by comparison to an adjustable loop device. Barrow et al similarly found that the ultimate load to failure of all 3 devices tested (fixed and adjustable loops) exceeded the forces likely to be experienced in a patient's knee during the early postoperative rehabilitation period. They also reported the adjustable loop devices lengthening to a clinically significant degree when subject to cyclic loading. However, they reported this lengthening significantly reduced for one adjustable loop device when the free suture ends were tied.

Barrow and Petre's papers examined loop strength and failure rates in a laboratory environment using a mechanical device for loop testing. Eguchi's work included testing loops fixed to porcine femurs and bovine femurs. Whilst recognised as models for such biomechanical testing, neither test scenario replicates the in-vivo situation that an ACL graft will face in human tissue.

The only clinical study comparing the loops was published by Boyle et al in 2015. In this retrospective study, the results of 188 patients were compared for 73 patients with an adjustable suspensory loop and 115 with a fixed loop. At varying time intervals of follow- up, no clinically statistically significant different outcomes were identified using stability testing via the KT1000 device and nor were differences found in graft failure. This study however, was not a prospective randomised study and has methodological flaws. In particular, there is a potential for bias in interpreting the assessment of the pivot shift and Lachman tests post-operatively as this was carried out by the operating surgeons who were not blinded to the type of surgery undertaken. Data was available for all 188 patients at the 6 month post-operative time frame- by which time graft healing should have occurred. However, only 58.5% of patients had data at 1 year follow-up and only 11.2% of patients achieved 2 year follow up. The graft diameter was statistically significantly larger in the adjustable loop cohort which can affect graft healing. Nevertheless, despite these limitations, this study outlined there was no detriment to using the adjustable loop system compared to the fixed loop in a clinical setting.

Thus the evidence of load to failure strength for all types of loop appears satisfactory, whilst some makes of adjustable loop appear to lengthen beyond acceptable levels in a laboratory situation after cyclic testing. We have carried out independent biomechanical testing of the loops being examined in this study and both met requirements for not lengthening excessively after cyclic loading and having pull to failure strength measurements in excess of those than would occur in daily life.

This clinical study therefore, aims to examine if there is any difference in clinical and functional outcome for patients undergoing ACL reconstruction using a hamstring autograft in a group of patients having a fixed length suspensory device used on the femoral side versus a group with an adjustable length one. It will be the first purely clinical prospective randomised study of these type of loops with the assessors of both clinical tests and the KT1000 device blinded as to which type of surgery the patient has undergone.

Methodology:

A randomised, prospective, study is to be set up to compare the results of 2 different ways of undertaking femoral fixation in ACL reconstruction surgery. One arm of the study will be randomised to have their surgery using a fixed length suspensory loop device for achieving femoral side graft fixation, and the other to have an adjustable suspensory loop used. The study will be carried out in the operating theatres, orthopaedic out-patients department and the physiotherapy department at the Royal Devon and Exeter (RD+E) Hospital.

Patients will be invited to take part in the study in one of 2 ways. Firstly, by their surgeon when they are initially listed for ACL reconstruction surgery at their out-patient consultation at the RD+E Hospital orthopaedic department. Alternatively, if they are identified from the current surgical waiting list as suitable for inclusion. In this latter case, they will be contacted by letter by their surgeon asking for permission for one of the research team to contact them to discuss the study. All participants will be sent a copy of the patient information leaflet. At their preparation for surgery appointment- usually 2-4 weeks before their operation, they will meet one of the research team who can answer any questions about the study. A study consent form will be signed at this meeting if the patient is willing to be involved in the research Patients who agree to enter the trial will be divided at random to enter the different treatment arms of the study. The randomization schedule will be determined using an on-line random assignment sequence generator (www.graphpad.com/quickcalcs/randomize1.cfm) and will be kept and controlled by the study co-ordinator, and the surgeons will not have access to this schedule. The randomisation details for each patient will be written on to a slip of paper and placed inside an opaque envelope. Each envelope is attributed to one patient and given a study number. One of the research team (study coordinator or research nurse) will supply the operating theatre staff with one of the envelopes containing the slip of paper upon which will be written the randomisation allocation for the patient undergoing surgery at that time. The operating theatre staff will inform the surgeon of the allocation. 150 patients will be initially included with allocation to either arm of the trial. The operating surgeon will not be able to read the slips before the envelope is opened, nor will they perform the randomisation which will be carried out by one of the investigators not carrying out the surgery on the individual patients i.e. the operating surgeon takes no part in the randomisation process.

Sample Size:

In 2015, at the RD+E Hospital 75 ACL reconstruction procedures were undertaken. 35 cases were performed at Sidmouth hospital giving a total of 110 per annum.

Lanzetti's paper (Ref 11) indicated that the mean and Standard Deviation (SD) values using the KT-1000 to measure Antero-Posterior (AP) translation of the tibia in relation to the femur were as follows:

Group a Group b KT 1000 Manual maximum 2.3+/-0.9 2.5+/-1 side to side difference (millimetres-mm) 2.1+/-1.2 2.3+/-1 Based on these values the study was powered to detect a Minimum Clinically Important difference (MCID) of 0.6 mm, which would shift the KT-1000 reading from 3.0 mm (upper bound of satisfactory level) to 3.6 mm (0.6 mm above the satisfactory upper bound).

Justification: If the true minimum difference (or Minimal Clinically Important Difference) between the experimental and control group KT-1000 measurement means is 0.6mm the researchers will need to recruit 60 cases in each group to be able to reject the null hypothesis that the population means are equal with probability (power) 0.9, type I error rate of 5% (significance) and mean SD of 1.0 (Lanzetti paper referred to above) An adjustment of 20% to account for drop outs would increase the number in each group to 75 and the total sample size to 150 cases.

Data Analysis:

Results of all the primary outcome between the 2 groups will be analysed at the 12 month time frames using students t-test to compare the groups. A stats package such as SPSS version 24 software will be used (SPSS Inc., Chicago, Illinois) for analysing the results.

Procedure:

Potential candidates for this study will be identified in one of 2 ways. Firstly, when patients are listed for ACL reconstruction surgery whilst attending orthopaedic out-patient clinics at the RD+E Hospital. At the time of this consultation they will be offered the opportunity to participate in the study. They will be given a copy of the information about the study and the consent form. They will have the opportunity therefore, to discuss the study with their family, friends or General Practitioner (GP) if they wish to do so. It will be explained that a member of the research team will contact them by telephone or letter to ask if they wish to participate in this research. Alternatively, patients will be identified from existing surgical waiting lists. In this case, they will be contacted by their surgeon in writing asking for their permission for one of the study team to approach them about the study. If permission is given, the patient will be sent a copy of the participant information sheet and a consent form so that they can decide if they would like to be involved. One of the research team- either the study coordinator or one of the research nurses- will then contact the patient and if they are willing to be involved, will obtain written consent for study participation. Consent is will be obtained at the preparation for surgery appointment which usually occurs 2-4 weeks before surgery.

3 copies of written consent will be obtained. One will be returned to the patient. One will be placed in the medical notes and one will be kept by the research team in the patient's case record file (CRF).

Patient Generated Clinical Outcomes/ Pre-operative Functional Assessment:

All ACL reconstruction patients attend the hospital for routine pre-operative assessment-whether involved in the study or not. At this appointment-usually 2-4 weeks before their operation- trial participants will complete the questionnaires related to the study: the Knee Osteo-arthritis Outcome Score (KOOS), the International Knee Documentation Committee (IKDC) subjective knee questionnaire, the Lysholm Knee Questionnaire and the Tegner activity score.

Initial Radiological Assessment:

Most patients will have undergone a Magnetic Resonance Image (MRI) scan of the affected knee prior to surgery as part of routine care. This test is not performed on all patients having this type of surgery, and is not one of the procedures being examined in this study; hence it is not necessary for every patient to undergo this.

Randomisation:

Randomisation will be to one of 2 arms of the study. The patient will either receive:

1. An ACL reconstruction using a fixed length suspensory loop for femoral fixation, or
2. An ACL reconstruction using an adjustable length suspensory loop for femoral fixation Tibial fixation for all participants will be as per routine care with an appropriately sized interference screw.

Patients who agree to enter the trial will be divided at random to enter the different treatment arms of the study. The randomization schedule will be determined using an on-line random assignment sequence generator (www.graphpad.com/quickcalcs/randomize1.cfm) and will be kept and controlled by the study co-ordinator, and the surgeons will not have access to this schedule. The randomisation details for each patient will be written on to a slip of paper and placed inside an opaque envelope. Each envelope is attributed to one patient and given a study number. One of the research team will supply the operating theatre staff with one of the envelopes containing the slip of paper upon which will be written the randomisation allocation for the patient undergoing surgery at that time. The operating surgeon will not be allowed to open the envelope. The patient will be assigned the study number and their randomisation slip returned to the study coordinator to be kept with the Masterfile copy of the consent form. A hand written note will be made by one of the research team in the orthopaedic section of the patient's medical notes after their surgery, confirming that they consented to the study and detailing which arm of the study they were allocated to.

Surgery:

Operating techniques will be standard ACL reconstruction techniques using hamstring autograft as used by the 2 surgeons involved in the study.

The operating surgeon will record in the operation note evidence of meniscal damage, cartilage and ACL status, including presence of any residual ACL.

Immediate Post-operative Care:

Patients will be discharged home allowed to fully weight-bear as comfort allows with walking aids for use for a 2 week period. They will be discharged wearing a locked knee brace. They will be reviewed at 2 days after surgery for a wound check and brace removal. They will be instructed in closed kinetic chain knee exercises, range of motion exercises, advised on cryotherapy and referred to the physiotherapy department for a formal ACL rehabilitation programme which will begin 2-3 weeks after surgery. This is all routine care in the researcher's institution.

Follow Up:

As per routine care, the patients will be followed up in the orthopaedic clinic at 2 and 6 weeks, 3 months, 6 months and 1 year post-operatively.

At the 6 month, 1 and 2 year timeframe they will repeat the KOOS, IKDC subjective knee score, Tegner Activity score and the Lysholm Knee questionnaire. These can be completed and posted from home by the patients or when they attend for KT1000 testing- see below.

Functional assessment using the KT1000 device will also be carried out at the 3 and 6 month and 1 year follow up time frames.

Physiotherapy will continue as clinical need dictates- as per routine care. If possible, all patients will undergo their rehabilitation at the RD+E Hospital to ensure standardisation of care. However, there will be practical logistical reasons why all patients will not be able to do this and they will have to have their physiotherapy in their local hospital.

Post-operative Radiological Assessment:

All participants will get a single Antero-Posterior (AP) and Lateral X-ray of the operated knee on the day of surgery as per routine care.

Data Storage The KOOS, IKDC subjective knee score, Tegner Activity Score and the Lysholm Knee Questionnaire are all undertaken by patients. This is in paper format and transcribed onto an Excel spread sheet on an RD+E Trust computer. The results of the KT1000 measurements will be also put on the spread sheet. The data will remain the property of the RD+E Hospital.

All of the remaining data associated with the study will be kept electronically on the hard drives of computers within the Exeter Knee Reconstruction Unit (EKRU). These are encrypted and password protected hospital computers. The data will only be accessible by members of the research team and the study sponsor who will need access for research regulatory purposes. The data will be analysed and reported.

The study Masterfile will be kept in the EKRU offices-an area that is inaccessible to the general public and for which staff require keypad door access.

Data Collation:

To be undertaken by the clinician undertaking the specific procedure concerned, the study coordinator or by research nurses attached to the Research and Development (R+D) department in the RD+E Hospital. The data will be stored on RD+E Hospital secure computers. Data will be entered into an Excel spread sheet for later transfer into a statistical package such as Statistical Package for the Social Sciences (SPSS) version 24 for analysis. All patient identifiers will be removed. The study data will be kept until the study analysis has been completed and then archived in accordance with the archiving Standard Operating Procedures (SOPs) of the study sponsor.

Data analysis:

Will be carried out by an appropriately qualified statistician.

Personnel:

* Chief Investigator-Andrew Toms (ADT)
* Surgeons-Vipul Mandalia (VIM) and Peter Schranz (PZS)
* Study coordinator-Patrick Hourigan (PGH)
* Functional outcome assessment team-Dean Chisling De Burgh (DCDB) -physiotherapy department RD+E Hospital.
* Database support provided by David Searle- surgical care practitioner in the EKRU.
* Clerical staff attached to the EKRU.

Confidentiality:

All of the research staff will be trained in guidelines for Good Clinical Practice (GCP) in research. All National Health Service (NHS) staff involved are bound by patient confidentiality requirements of the NHS.

The study participants General Practitioner (GP) will be informed that their patient is involved in the research- particularly as the patient may wish to discuss their involvement in the research with their GP.

All of the data associated with the study will be kept electronically on the hard drives of computers within the Exeter Knee Reconstruction Unit (EKRU). It will be stored on encrypted and password protected hospital computers. The data will only be accessible by members of the research team and by the R+D department at the RD+E Hospital who will require access to the data to ensure compliance with the protocol.

When the data is to be sent to the statistician for analysis, it will be anonymised and only a study number used for identification. The statistician uses password and encrypted computers.

At the end of the study (see timescales below), all research data will be archived in line with the sponsors SOPS. Radiographs and scans will remain on the secure hospital systems as per routine care.

Timescales:

Approximately 110 ACL reconstructions carried out per annum by the surgeons within the research team. Allowing 50% declining recruitment, not meeting entry criteria or missed for logistical reasons this will leave 55 potential participants per annum. Thus recruitment should be in approximately 2 years and 8 months. Follow up is for 2 years post entry into the study as outlined above.

It will take a further 1 year for data analysis, project write up and submission for publication post study end.

Study data will be archived as per the study sponsors archiving SOP's after completion of the study.

Dissemination of Results:

The participants will be informed in writing of the results if they so desire. The R+D department at the RD+E will be informed of the results.

The research team plan to present the results both nationally and internationally at knee surgery conferences and to publish the results in a peer reviewed journal.

The team will also present the results to the 2 patient networks in Exeter: The Patient Research Panel and The Patient Knee Support Group

Impact of Results:

The impact of this study as yet is unknown. If the research identifies a clear advantage of one study arm over the others, then it is likely that this technique will become the standard ACL reconstruction procedure within the RD+E Hospital- with the aim of providing patients with the best clinical and functional results after their ACL reconstruction surgery. Similarly, if a clear difference is found in one study arm, one would hope that presentation of the results to colleagues at other institutions will result in better long term results for their patients.

In the event that no technique proves superior to the others, then this will provide surgeons with the reassurance that no matter what their preferred technique, their patient is not being disadvantaged.

If results between both arms of the study are the same, there is a potential cost saving for the NHS if only one size of adjustable suspensory loop needs to be kept in stock a opposed to multiple different sizes of the fixed loop device.

Conflicts of Interest:

The Exeter Knee Reconstruction Unit has received external funding to allow them to undertake studies as this. This is subject to a Masters Service Agreement (MSA) and the monies are already in place.

Both devices being studied are made by the same company and thus using one or the other is of no financial benefit to the manufacturer.

ADT and VIM undertake consultancy work for Stryker UK and will complete the necessary paperwork for this.

Patient Involvement:

The research team have consulted with patients on the feasibility of participating in the study at all and in particular about the demands of attending the appointments for functional assessment. The commitment for the majority of the study is the same whether patients are involved in the research or not but nevertheless the research team will emphasise the need for attendance. However, rehabilitation for patients living in Exeter is undertaken at the RD+E site. For some patients who live in the surrounding areas, rehabilitation could normally be undertaken in their local community hospital using current protocols. Ideally the research team would like all patients to attend for rehabilitation at the RD+E so as to standardise care. However, this will not always be possible as patients may have logistical difficulty travelling to Exeter when the study population is drawn from a wide geographical area. If patients do not wish or cannot travel to Exeter for this however, they will have to come to Exeter on 3 extra separate occasions for the KT100 functional test. Attendance at all time frames is critical for completion of the functional outcome assessment. This is both the study primary outcome measure but also the safety net of ensuring neither study arm is failing catastrophically. It was stressed by the patient representatives that the patients need to be fully informed of the commitment required should they agree to take part.

The research team have consulted on the design and wording of the patient information leaflet and the consent form. Various changes were recommended in particular to the patient information leaflet- all were implemented.

Risks of the Study:

The research team do not believe involvement in this study changes the risks from surgery that the patients already face as a part of routine care.

Monitoring Adverse Events/Stopping the Study:

A log of adverse events will be kept by the study coordinator. Adverse events occurring in the immediate peri and post-operative events should be reported to the coordinator by the consultant surgeon in charge of the case. Adverse events may be identified in clinic and again, the surgeon concerned should report these back to the coordinator to be logged and further action considered if necessary after discussion with the study sponsor.

It is possible that adverse events will occur that are dealt with either by the Accident and Emergency (A+E) department, the patient's GP or other hospitals. These may not be readily apparent to the research team. The research team will therefore specifically ask participants to inform their surgeon if any complications or adverse events occur and similarly ask the surgeons to specifically ask their patients for this information at each clinic attendance.

A meeting of the research team will be held on a 3 monthly basis to discuss progress of the study, any specific problems and to consider whether there are any justifications for stopping the study. As both techniques being studied of performing ACL are already part of routine practice, the research team do not anticipate identifying an unexpected complication that would necessitation an early termination of the study.

Ethical Approval:

Ethical approval for this study will be sought from the National Research Ethics Committee via the Health Research Authority.

ELIGIBILITY:
Inclusion Criteria:

* Isolated ACL deficient knee without other ligament injury
* Patients who have a small meniscal tear that requires flap excision during the ACL surgery can be included in the study-see exclusion criteria below.
* Patient has signed an ethics committee approved consent form
* Surgery to be performed at either at The Royal Devon and Exeter Hospital or Sidmouth Hospital.
* Patient is willing and able to comply with postoperative scheduled clinical and functional evaluations and rehabilitation
* Patients undergoing ACL reconstruction using hamstring autograft

Exclusion Criteria:

* Patients <16 years old
* Refusal to consent to participate in the study
* Previous knee surgery or serious knee injuries in the operative knee
* Obvious clinical knee malalignment-i.e. visible on clinical examination
* Multi ligament knee injuries.
* Moderate to severe degenerative changes present within the knee joint.
* If a simultaneous sub-total meniscectomy involving 50% or more of the meniscus has to be performed
* Patients who also have a postero-lateral corner injury
* Patient has a neuromuscular or neurosensory deficiency
* Pregnancy

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The assessment of knee joint stability via a comparison of left and right sided anterior tibial translation | 12 months after surgery
  Anterior tibial translation will be assessed using the KT1000 device using a students t-test or a non-parametric equivalent if the data is not normally distributed e.g. the Mann- Whitney u test to compare the groups. The Minimal Clinically Important Difference between the groups will be 0.6mm above the acceptable threshold of 3mm

SECONDARY OUTCOMES:
An assessment of Functional outcome (1) using the results of the Knee Osteo-Arthritis Outcome Score (KOOS) | 6 months after surgery
  The secondary outcome measures (KOOS) data results will be evaluated using the same t-test or Mann- Whitney u test at the 6 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
An assessment of Functional outcome (2) using the results of the Knee Osteo-Arthritis Outcome Score (KOOS) | 12 months after surgery
  The secondary outcome measures (KOOS) data results will be evaluated using the same t-test or Mann- Whitney u test at the 12 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
An assessment of Functional outcome (3) using the results of the Knee Osteo-Arthritis Outcome Score (KOOS) | 24 months after surgery
  The secondary outcome measures (KOOS) data results will be evaluated using the same t-test or Mann- Whitney u test at the 24 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
An assessment of Functional outcome (4) using the results of the International Knee Documentation Committee (IKDC) subjective questionnaire | 6 months after surgery
  The secondary outcome measure (IKDC) data results will be evaluated using the same t-test or Mann- Whitney u test at the 6 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
IKDC subjective knee questionnaire | 12 months after surgery
  The secondary outcome measure (IKDC) data results will be evaluated using the same t-test or Mann- Whitney u test at the 12 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
IKDC subjective knee questionnaire | 24 months after surgery
  The secondary outcome measure (IKDC) data results will be evaluated using the same t-test or Mann- Whitney u test at the 24 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
Lysholm knee score: Functional outcome 7 | 6 months after surgery
  The secondary outcome measure (Lysholm Knee Score) data results will be evaluated using the same t-test or Mann- Whitney u test at the 6 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
Lysholm knee score: Functional outcome 8 | 12 months after surgery
  The secondary outcome measure (Lysholm Knee Score) data results will be evaluated using the same t-test or Mann- Whitney u test at the 12 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
Lysholm knee score: Functional outcome 9 | 24 months after surgery
  The secondary outcome measure (Lysholm Knee Score) data results will be evaluated using the same t-test or Mann- Whitney u test at the 24 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
Tegner activity scale: Functional outcome 10 | 6 months after surgery
  The secondary outcome measure (Tegner Activity Scale) data results will be evaluated using the same t-test or Mann- Whitney u test at the 6 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
Tegner activity scale: Functional outcome 11 | 12 months after surgery
  The secondary outcome measure (Tegner Activity Scale) data results will be evaluated using the same t-test or Mann- Whitney u test at the 12 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.
Tegner activity scale: Functional outcome 13 | 24 months after surgery
  The secondary outcome measure (Tegner Activity Scale) data results will be evaluated using the same t-test or Mann- Whitney u test at the 24 month timeframe. If the secondary outcome data shows sufficient power and allows it, we will analyse the secondary outcomes at the other timeframes using repeated measures of ANOVA.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Toms, MSc FRCS, Principal Investigator — RD+E Hospital NHSFT
Locations (1):
- Royal Devon and Exeter Hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
we do not plan to give the data to others